CLINICAL TRIAL: NCT00234598
Title: Oral Care Intervention in Mechanically Ventilated Adults
Brief Title: Strategies to Prevent Pneumonia (SToP Pneumonia)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: VCU1006; R01NR007652 (NIH); R01 NR07652 (NIH)
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Pneumonia; Dental Health; Critical Care
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pneumonia | interventions — Toothbrushing; Chlorhexidine

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control group, usual care (No Intervention): Usual care with no study interventions provided; no tooth brushing intervention and no chlorhexidine intervention. Usual care
- Tooth brushing only (Active Comparator): Tooth brushing by study personnel three times per 24 hours (TID) without chlorhexidine application.
  Interventions: Procedure: Toothbrushing only
- Chlorhexidine only (Active Comparator): Oral application of chlorhexidine 0.12% oral solution twice per 24 hours (BID) without tooth brushing.
  Interventions: Procedure: Chlorhexidine only
- Toothbrushing and chlorhexidine (Active Comparator): Tooth brushing by study personnel three times per 24 hours (TID) and oral application of chlorhexidine 0.12% oral solution twice per 24 hours (BID)
  Interventions: Procedure: Toothbrushing and Chlorhexidine

INTERVENTIONS:
Procedure: Toothbrushing only — Toothbrushing three times per 24 hours without chlorhexidine
  Arms: Tooth brushing only
Procedure: Chlorhexidine only — Chlorhexidine oral rinse twice per 24 hours without toothbrushing
  Arms: Chlorhexidine only
Procedure: Toothbrushing and Chlorhexidine — Toothbrushing three times per 24 hours plus chlorhexidine twice per 24 hours.
  Arms: Toothbrushing and chlorhexidine

SUMMARY:
This study tests whether special oral care provided by nurses to critically ill patients who are on a breathing machine (mechanical ventilator) can help to reduce the build-up of dental plaque on the teeth and reduce the risk of pneumonia.

DETAILED DESCRIPTION:
Pneumonia is the leading cause of death from hospital-acquired infections. Intubation and mechanical ventilation greatly increase the risk of bacterial ventilator associated pneumonia. Growth of potentially pathogenic bacteria in dental plaque of critically ill patients provides a nidus of infection for microorganisms that have been shown to be responsible for the development of Ventilator Associated Pneumonia. Since these organisms are concentrated in dental plaque, removal of organisms from the oral cavity by oral care interventions is a theoretically attractive method to reduce the risk of development of Ventilator Associated Pneumonia. However, evidence-based protocols for oral care of mechanically ventilated patients are not available. Results of the study have the potential to improve nursing care, and to positively affect patient well-being, morbidity, mortality, and health care costs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, admitted to one of four intensive care units at the study hospital, breathing tube in place, and on a breathing machine (mechanical ventilator)

Exclusion Criteria:

* Breathing tube in place for more than 24 hours prior to entry into the study, absence of teeth, or a medical diagnosis of pneumonia when the breathing tube is put in.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2002-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Reduction of build-up of dental plaque on the teeth and reduced risk of pneumonia in critical care patients, as a result of special oral care provided by nurses. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Munro, RN, ANP,PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States